CLINICAL TRIAL: NCT00974129
Title: Infantile Hemangioma Tumor Size and C/T Polymorphism Within CTCF Binding Site Six
Brief Title: A Study of CCCTC-binding Factor (CTCF) in Infantile Hemangiomas
Status: Withdrawn | Type: Observational
Why Stopped: no subjects were enrolled, study was halted due to study staff departure
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 0507000430; Yale-0430
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Hemangioma
MeSH Terms: conditions — Hemangioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Over the course of the study, one blood draw will be performed on each patient. This blood will be used for genetic analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with Infantile Hemangiomas

SUMMARY:
The purpose of this study is to evaluate the genotype of CTCF, a proven transcription factor, in patients with infantile hemangiomas and to monitor tumor growth. The investigators aim to determine whether or not the CTCF genotype might serve as an early and reliable predictor of tumor growth.

DETAILED DESCRIPTION:
This study seeks to examine a potential relationship between CTCF genotype and hemangioma size and growth rate. In addition to the initial visit, patients will return to our clinic for evaluation at two weeks, one month, two months, six months, and one year. At each visit, patients' hemangiomas will be measured and photographed. At one point over the course of evaluation, a blood sample will be taken from each patient for evaluation of C/T polymorphism at CTCF binding site six.

ELIGIBILITY:
Inclusion Criteria:

* Hemangioma must appear within one month prior to enrollment

Exclusion Criteria:

* Hemangioma appeared before one month prior to enrollment

Max Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients to be recruited will include infants with hemangiomas on any part of their body.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Narayan, MD, Principal Investigator — Yale University
Locations (1):
- Yale Dermatology Associates, New Haven, Connecticut, United States